CLINICAL TRIAL: NCT05698758
Title: A Randomized Controlled Trial of Intranasal Dexmedetomidine for Adult Patients Undergoing Phacoemulsification Cataract Surgery
Brief Title: Intranasal Dexmedetomidine for Adult Patients Undergoing Phacoemulsification Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Yuehong Zhang, Clinical Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-2022-160-01
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Preoperative Sedation
Keywords: Cataract; Preoperative sedation; Dextromethoridine; Patient satisfaction
MeSH Terms: conditions — Cataract; Patient Satisfaction | interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dextrometropine group (Experimental): Approximately 45 - 60 minutes before cataract surgery, patients in the dextrometropine group were given dextrometropine (1.0μg.kg-1).
  Interventions: Drug: Dextrometropine and 0.9% sodium chloride solution
- placebo group (Placebo Comparator): Approximately 45 - 60 minutes before cataract surgery, patients in the placebo group were given 0.9% sodium chloride solution (1.0μg.kg-1).
  Interventions: Drug: Dextrometropine and 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Dextrometropine and 0.9% sodium chloride solution — Intranasal dexmedetomidine or 0.9% sodium chloride solution as a sedative premedication for patients undergoing cataract surgery
  Other Names: Dexmedetomidine Hydrochloride

SUMMARY:
The investigators designed this study to examine whether the intranasal dexmedetomidine, as a preoperative drug, could improve the satisfaction of adult patients undergoing phacoemulsification cataract surgery.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized controlled study. Patients over 65 years old were selected for phacoemulsification combined with intraocular lens implantation under topical anesthesia. Participants were randomly divided into two groups: dextrometropine group and placebo group, and were masked until the end of this study. Approximately 45 - 60 minutes before surface anesthesia, patients in the dextrometropine group were given dextrometropine (1.0μg.kg-1), patients in the placebo group were given the same amount of saline. The primary end point of this study is the patient satisfaction. Patient satisfaction was assessed using a 3-point satisfaction score on a scale. Anxiety of perioperative patients was assessed using a 4-point anxiety score on a scale. Secondary endpoints include blood pressure, heart rate, blood oxygen saturation, operation time, operative complications and adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria: Cataract patients over 65 years scheduled for elective phacoemulsification and intraocular lens implantation in Department of Ophthalmology, Guangzhou First People's Hospital will be recruited in this study. Recruited patients shall own normal intelligence and understanding capability and their best corrected visual acuity more than 0.1 in either eye.

Exclusion Criteria: 1) a known allergy or hypersensitivity to dextrometropine or other anesthetics; 2) a previous history of heart disease; 3) a heart rate (HR) <45 beats per minute (bpm); 4) a second- or third-degree atrioventricular block; 5) patients on antihypertensive drugs, such as α-methyldopa, clonidine, or other α2-adrenergic agonists; 6) asthma; 7) sleep apnea syndrome; 8) organ dysfunction; 9) patients with mental illness; and 10) the long-term use of sedatives and analgesics.

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall patients satisfaction with preoperative sedation | Operation day
  Patient satisfaction was assessed using a 3-point satisfaction score on a scale (1 = highly satisfactory, 2 = acceptable, and 3 = unacceptable). The minimum value is 1 and maximum is 3. Higher scores mean a worse outcome.
Anxiety of perioperative patients | Operation day
  Anxiety of perioperative patients was assessed using a 4-point anxiety score (1 = combative, 2 = anxious, 3 = calm, and 4 = amiable). The minimum value is 1 and maximum is 4. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Effects of preoperative sedation on patients' vital signs and operation time | Perioperative period
  Blood pressure, heart rate, blood oxygen saturation, operation time, operative complications and adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Zhang, PhD, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No